CLINICAL TRIAL: NCT00007943
Title: A Phase II Study Of Twenty-Four Hour Infusion Gemcitabine For Advanced Colorectal Cancer
Brief Title: Gemcitabine in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: REBACDR0000068355; CCCWFU-59198; NCI-914
Record Dates: First submitted 2001-01-06; First posted 2004-04-13 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine in treating patients who have advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with advanced colorectal cancer treated with gemcitabine.
* Determine the toxic effects of this drug in these patients.
* Determine the progression-free survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV continuously over 24 hours on days 1, 8, and 15. Treatment repeats every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 12-41 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced colorectal cancer that has failed at least 1

prior course of fluoropyrimidine-based chemotherapy

Measurable and/or evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* ALT and/or AST no greater than 3 times ULN (no greater than 10 times ULN if
* secondary to hepatic involvement by tumor

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No history of cardiac arrhythmias requiring chronic treatment beyond an
* acute event (e.g., arrhythmias during severe electrolyte abnormalities
* allowed)
* No active cardiac disease requiring treatment other than hypertension,
* stable angina, or chronic valvular disease

Other:

* No other malignancy within the past 5 years except curatively treated
* (including surgically cured) cancer
* No serious medical or psychiatric illness that would preclude study
* No active uncontrolled bacterial, fungal, or viral infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 3 prior chemotherapy regimens
* Must have 1 prior fluorouracil-based regimen and 1 other cytotoxic agent
* (e.g., irinotecan)
* More than 4 weeks since prior chemotherapy
* Prior gemcitabine allowed
* No other concurrent antineoplastic therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* More than 4 weeks since prior radiotherapy

Surgery:

* More than 4 weeks since prior surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2000-09-01 (Actual); Primary Completion 2001-02-27 (Actual); Study Completion 2001-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Savage, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States